CLINICAL TRIAL: NCT06738615
Title: Assessing the Impact of Diastolic Dysfunction on the Presence of Symptoms in Patients with Primary Mitral Regurgitation.
Brief Title: Assessing the Relationship Between Symptoms and Mitral Regurgitnant. Severity
Status: Recruiting | Type: Observational
Sponsor: Atlantic Health System (Other)
Responsible Party: Principal Investigator, Seth Uretsky, Medical Director, Cardiovascular Imaging, Atlantic Health System
Other Study IDs: 2223778
Record Dates: First submitted 2024-12-08; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Mitral Insufficiency
Keywords: mitral regurgitation; symptoms; exercise capacity
MeSH Terms: conditions — Mitral Valve Insufficiency | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Mitral Regurgitation: Patients with mitral regurgitation undergoing a left heart catheterization prior to mitral valve surgery or mitral valve clip.
  Interventions: Diagnostic Test: Pressure volume loop evaluation; Diagnostic Test: cardiovascular magnetic resonance imaging; Diagnostic Test: Cardiopulmonary exercise testing (CPET); Diagnostic Test: Kansas City Cardiomyopathy Questionairre

INTERVENTIONS:
Diagnostic Test: Pressure volume loop evaluation — During the left heart catheterization there are catheters which are introduced into the left ventricle to measure left ventricular pressures and into the coronary arteries to assess their patency. This study will require the placement of an additional specialized catheter made into the left ventricle to measure the change of pressure and volume during the cardiac cycle. This will allow the measurement of heart muscle stiffness.
Diagnostic Test: cardiovascular magnetic resonance imaging — Patients will undergo standard cardiovascular magnetic resonance imaging of their heart to measure their heart size, heart function, and severity of mitral regurgitation. In addition, contrast will be administered and heart tissue will be assessed for scarring or fibrosis.
Diagnostic Test: Cardiopulmonary exercise testing (CPET) — A CPET will be performed to objectively measure a patient ability to perform exercise.
Diagnostic Test: Kansas City Cardiomyopathy Questionairre — This is a short questionnaire which objectively quantifies symptom burden

SUMMARY:
The current American College of Cardiology/American Heart Association (ACC/AHA) guidelines recommend surgery in patient with mitral regurgitation (MR) based on 1) the severity of MR and 2) the presence or absence of symptoms. Studies have shown that Cardiovascular Magnetic Resonance (CMR) is an accurate method to quantify the severity of MR. However, studies have also shown that symptoms are not necessarily related to the presence of symptoms. Thus, there appears to be a disconnect between the severity of MR and symptoms. Recent analysis of our data has shown that females and older patients with smaller ventricles, lower stroke volumes, and lower regurgitant volume relative to regurgitant fraction tend to be symptomatic. These findings suggest that decreased left ventricular compliance, i.e. diastolic dysfunction, may play an important role as an etiology of symptoms in patients with mitral regurgitation. The aim of this study is to study the presence of diastolic dysfunction in patients with MR and its association with symptom burden and exercise capacity.

DETAILED DESCRIPTION:
The study is an observational study of patients with mitral regurgitation undergoing LHC prior to mitral valve surgery or percutaneous mitral valve intervention. Prior to patients LHC they will undergo testing using CMR, CPET, and KCCQ. During the LHC, patients will undergo evaluation of intracardiac pressures and volumes using a specialized catheter which measures pressure and volume changes throughout the cardiac cycle.

CMR- CMR evaluation will quantify mitral regurgitant volume and fraction, right and left atrial size and function, and myocardial scar quantification.

CPET- objectively assess patients exercise capacity. KCCQ- is a standard questionnaire designed to assesses patients quality of life and symptom burden.

LHC- Pressure-volume loops will be measured during LHC. This will quantify left ventricular compliance and assess patients for the presence of diastolic dysfunction.

These evaluations will help us better understand the relationship between symptoms, exercise capacity, severity of MR and diastolic dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years of age
* Able to give informed consent
* Primary (degenerative) mitral regurgitation
* LVEF >=50%
* Undergoing cardiac catheterization
* Able to exercise on a treadmill

Exclusion Criteria:

* Unable to give informed consent
* Secondary (functional) mitral regurgitation
* LVEF <50%
* Known coronary artery stenosis >=70% or past revascularization
* More than mild aortic stenosis, mitral stenosis, aortic regurgitation, tricuspid regurgitation, or pulmonic regurgitation
* Hypertrophic cardiomyopathy
* Pregnancy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study if for patients with mitral regurgitation who are undergoing cardiac catheterization prior to mitral valve surgery or mitral valve clip.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-01-02 (Estimated); Primary Completion 2027-01-02 (Estimated); Study Completion 2027-05-02 (Estimated)

PRIMARY OUTCOMES:
Diastolic Dysfunction Symptoms/exercise capacity | Enrollment to testing completed 8 weeks
  Assess the relationship between diastolic dysfunction. Diastolic dysfunction is measured by pressure volume loop assessment. Diastolic disfunction will be compared to patients symptom burden (as quantified by KCCQ) and exercise capacity (as quantified by CPET).

SECONDARY OUTCOMES:
Mitral regurgitation severity and measures of diastolic dysfunction | enrollment to 8 weeks
  MR volume and fraction compared to diastolic dysfunction as measured by pressure volume loop assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Morristown Medical Center, Morristown, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided